CLINICAL TRIAL: NCT06582901
Title: Cognitive Training vs. Treatment as Usual to Improve Functioning and Reduce Transition Rates in Tunisian CHR Youth: A Feasibility Study
Brief Title: Interventions for Clinical High Risk Youth in Tunisia
Acronym: CHRTUNISIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ventura, Joseph, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#23-001029; R21MH131319 (NIH)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Clinical High Risk for Psychosis (CHR)
Keywords: clinical High Risk youth; cognitive training; enhanced treatment as usual; transition to psychosis
MeSH Terms: interventions — Cognitive Training; Models, Biological

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial (RCT) study that is comparing two interventions: one is experimental and involves computer-based cognitive training using HappyNeuron and the Neuropsychological Educational Approach to Cognitive Remediation (CT-NEAR) model vs Enhanced Treatment as Usual (E-TAU).
Who Masked: Outcomes Assessor
Masking Description: One clinical rater will be unaware of the treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Computer Based Cognitive Training (CT) Programs delivered in a group setting using the Neuropsychological Educational Approach to Cognitive Remediation (NEAR) model.
  Interventions: Behavioral: Cognitive training (CT) plus the neuropsychological educational approach to cognitive remediation (NEAR) model and an Enhanced - Treatment as Usual (E-TAU)
- Enhanced Treatment as Usual (Active Comparator): Enhanced Treatment as Usual (E-TAU) sessions are delivered in a group therapy format and guided by the principles of Cognitive Behavioral Therapy (CBT). The E-TAU sessions focus on helping individuals identify and change negative thought patterns and behaviors that contribute to emotional distress and mental health issues.
  Interventions: Behavioral: Enhanced - Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive training (CT) plus the neuropsychological educational approach to cognitive remediation (NEAR) model and an Enhanced - Treatment as Usual (E-TAU) — Psychosocial interactions computer-based cognitive training (CT) administered in a group setting that includes the Neuropsychological Educational Approach to Cognitive Remediation (NEAR) model:
  Arms: Cognitive Training
Behavioral: Enhanced - Treatment as Usual — The Enhanced-Treatment as Usual (E-TAU) sessions are delivered in a group therapy format and guided by the principles of Cognitive Behavioral Therapy (CBT). Participants learn to develop coping skills and are educated on how to improve distortions to reduce anxiety and depression.
  Arms: Enhanced Treatment as Usual

SUMMARY:
Study participants will take part in one of the two types of treatments aimed at improving daily functioning as follows: either a Cognitive Training (CT) Program or an Enhanced - Treatment as Usual (E-TAU) Group. All group treatments will be provided at Razi Hospital and one of the sessions will be conducted at home. The Cognitive (thinking skills) Training and Neuropsychological Education Approach to Remediation (CT-NEAR) is a form of cognitive (thinking skills) training that consists of computer-game like brain exercises, learning about thinking skills strategies, and a "bridging group" to help participants use what is learned in daily life. Cognitive exercises are generally fun and playful and are done on a computer. The aim is to train thinking skills and ability to function better in daily life such as at school, university, or at work, or with friends and family. The program lasts 12 weeks with two weekly sessions in groups of 3 to 4 participants. Each session is 1½ hours in length and one of the sessions is which lasts 30 minutes is conducted at home using a tablet that will be provided by the study investigators.

DETAILED DESCRIPTION:
RESEARCH STRATEGY Recruitment of Study Participants Potential study participants are help-seeking youth recruited through the network of trained mental health professionals at schools and universities of the Greater Tunis area (see above) as well as through the CHiRP network at the outpatient departments of Razi University Hospital and Mongi Slim University Hospital.

Randomization to Cognitive Training (CT-NEAR) vs. Enhanced Treatment as Usual (E-TAU) After study entry, patients will be randomized to Cognitive Training (CT-NEAR) or Enhanced Treatment as Usual (E-TAU) using a 1:1 randomization immediately after completion of the baseline assessment battery. Both treatments will last 3 months. Participants in the two conditions will receive treatment which will be carefully tracked and all medication types and doses recorded. The conditions will be matched on all key variables such as amount of therapist and in-clinic time by offering group activities for participants in the E-TAU condition. A clinical and neurocognitive assessment battery will be administered to all participants at baseline by masked assessors. The clinical assessments (symptoms and functioning) will be repeated at 6 weeks (mid-point), and the full assessment battery will be repeated at the 3-month conclusion of the randomized treatment. We will examine the effects of the treatment on neurocognitive functioning, conversion, and role and social functioning.

Cognitive Training Using the Neuropsychological Education Approach to Remediation (CT-NEAR) Enhanced Treatment as Usual Comparison Group The E-TAU condition will consist of regular contact with mental health professionals in the outpatient clinic which involves conducting and monitoring of psychosocial interventions such as Cognitive Behavior Therapy groups for depression and anxiety, case management, supportive counselling, a psychoeducation group, and watching films at home for 30 minutes on a tablet. None of these interventions target improvement in cognition. Participants in the E-TAU condition will receive all of the baseline and follow-up clinical and neurocognitive assessments. The E-TAU condition will be matched for therapist time, group interaction time, and the use of a tablet at home. After the 3-month E-TAU period, participants will be offered participation in the cognitive training and will of course not be included in the CT-NEAR study sample.

Implementation of the Intervention Alignment with National Institute of Mental Health (NIMH) Strategic Plan: The current proposal aligns with several components of the NIMH Strategic Plan 2020.

ELIGIBILITY:
Inclusion Criteria:

* Meets Comprehensive Assessment for At Risk Mental States (CAARMS) criteria for Clinical High Risk
* If under the age of 18, the subject has a parent or guardian who can sign consent forms
* Premorbid Intelligence Quotient not less than 70
* Sufficient fluency in Arabic, French, or English to avoid invalidating research measures
* Residence likely within commuting distance of Razi University Hospital

Exclusion Criteria:

* Evidence of known neurological disorder, e.g. epilepsy or significant head injury that could account for the CHR symptoms
* Evidence of significant and habitual alcohol or substance use in the 6 months prior to study entry
* Evidence that the clinical high-risk symptoms were substance-induced

Ages: 14 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Functioning | Baseline, 3 months
  Neurocognitive Test Battery. Scored on a composite of various cognitive tests will indicate improved, not improved at follow-up. The composite score ranges from 0 to 50 with higher scores indicating greater improvement.

SECONDARY OUTCOMES:
Global Functioning Scale - Role and Social | Baseline, 3 months
  Interview-based assessment of work or school functioning and of social functioning. Scores range from 0-100 with higher score indicating better functioning.
Comprehensive Assessment of At-Risk Mental States | Baseline, 3 months
  Interview based assessment of clinical status assess change in clinical status from baseline to post - intervention. The scores range from 0-60 with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ventura, Ph.D., Principal Investigator — UCLA Department of Psychiatry & Biobehavioral Sciences
Locations (1):
- Razi University Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No